CLINICAL TRIAL: NCT01606904
Title: The Effect of CBT- Based Weight Loss Program on Eating Behavior, Weight Loss Result and Risk for Coronary Heart Diseases and Type 2 Diabetes
Brief Title: The Effect of CBT- Based Weight Loss Program on Obesity
Acronym: CognObe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Juho Vainio Foundation (Other); Yrjo Jahnsson Foundation (Other); Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Anna-Maria Keränen, P.h.D, clinical nutritionist, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 58/2012
Record Dates: First submitted 2012-05-21; First posted 2012-05-28 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Obesity; Hypercholesterolemia; Diabetes Mellitus, Type 2; Anhedonia
MeSH Terms: conditions — Obesity; Hypercholesterolemia; Diabetes Mellitus, Type 2; Anhedonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weight loss counseling (Experimental): Cognitive behavioral therapy - based weight loss program
  Interventions: Behavioral: Cognitive behavioral therapy -based weight loss program
- Control (Other): Short term weight loss counseling, control group
  Interventions: Behavioral: Cognitive behavioral therapy -based weight loss program

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy -based weight loss program — CBT-based program includes 20 group visits

SUMMARY:
The investigators purpose is to study how CBT (cognitive behavioral therapy)-based weight loss program affects on eating behavior, weight loss and risk factors for CHD (coronary heart diseases)and type 2 diabetes. Moreover, the investigators aim is to recognize subjects suffering from anhedonia (one of the core symptoms of depression, lack of pleasure) and follow how they benefit from the program in order to achieve maintained weight loss. Also, the associations between weight loss, physical activity and musculoskeletal disorders are studied.

DETAILED DESCRIPTION:
Obesity is an increasing problem and effective weight loss methods are needed. The study is randomized follow-up study with 9 months intervention and three (3) years follow-up period. The study is organized in Oulu University Hospital, Department of Internal Medicine. Eighty (80)obese, 20-65 years, study subjects will be randomized into intervention or control group.

The hypothesis of the CognObe study is: CBT (cognitive behavioral therapy)-based weight loss program is successful in sustained and favourable change in eating behavior and weight as well as decreased risk for coronary heart diseases or type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30

Exclusion Criteria:

* other concurrent weight loss programs
* disease which prevents weight loss
* medication which affects on weight loss

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
change in weight | baseline, 9 months, 1,2 and 3 years
  kilograms

SECONDARY OUTCOMES:
change in eating behavior | baseline, 9 months, 1,2 and 3 years
  emotional eating, uncontrolled eating, cognitive restraint, binge eating symptoms
change in total cholesterol,HDL, LDL,Trigly and glucose | baseline, 1,2 and 3 years
  change in laboratory values
DNA | baseline
  for genetic analyses
change in incretins | baseline, 12, 24 and 36 months
  change in incretins

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Maria Teeriniemi (nee Keränen), Principal Investigator — Oulun University Hospital
Locations (1):
- Deparment of Internal Medicine, Oulu University Hospital, Oulu, Finland

REFERENCES:
- [Background] Keranen AM, Savolainen MJ, Reponen AH, Kujari ML, Lindeman SM, Bloigu RS, Laitinen JH. The effect of eating behavior on weight loss and maintenance during a lifestyle intervention. Prev Med. 2009 Aug;49(1):32-8. doi: 10.1016/j.ypmed.2009.04.011. Epub 2009 May 4. PMID 19406146
- [Background] Keranen AM, Strengell K, Savolainen MJ, Laitinen JH. Effect of weight loss intervention on the association between eating behaviour measured by TFEQ-18 and dietary intake in adults. Appetite. 2011 Feb;56(1):156-62. doi: 10.1016/j.appet.2010.10.004. Epub 2010 Oct 16. PMID 20955744
- [Background] Keranen AM, Rasinaho E, Hakko H, Savolainen M, Lindeman S. Eating behavior in obese and overweight persons with and without anhedonia. Appetite. 2010 Dec;55(3):726-9. doi: 10.1016/j.appet.2010.08.012. Epub 2010 Aug 27. PMID 20801180